CLINICAL TRIAL: NCT05398185
Title: WiseApp for Spanish-Speaking Latino Persons Living With HIV (PLWH) in the United States (US) and the Dominican Republic (DR)
Brief Title: WiseApp for Spanish Speakers Living With HIV
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Clínica de Familia La Romana, Dominican Republic (Unknown)
Responsible Party: Principal Investigator, Rebecca Schnall, RN, MPH, PhD, Mary Dickey Lindsay Professor of Disease Prevention and Health Promotion, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: AAAT8632; 1R18HS028523-01 (AHRQ)
Record Dates: First submitted 2022-05-25; First posted 2022-05-31 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: HIV Infections; Acquired Immune Deficiency Syndrome; Sexually Transmitted Diseases, Viral
Keywords: People living with HIV (PLWH); Antiretroviral therapy (ART); Mobile Health; Spanish Speakers; Latinos
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; Sexually Transmitted Diseases, Viral

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants will be randomly assigned to one of two trial arms using sequentially numbered, opaque, sealed envelopes containing the intervention assignment, which the staff member opens at the moment of randomization
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Control (No Intervention): The control includes standard health services offered at each site (e.g., mental health services, case-management, referral to clinical care) and a brief adherence educational session.
- Intervention (Experimental): Participants randomized to intervention will receive the CleverCap pill bottle, an innovative technology that dispenses only the prescribed amount of medication, keeps track of medications dispensed, and communicates wirelessly with the WiseApp.
  Interventions: Device: CleverCap

INTERVENTIONS:
Device: CleverCap — The CleverCap pill bottle is an innovative technology that dispenses only the prescribed amount of medication, keeps track of medications dispensed, and communicates wirelessly with the WiseApp to deliver medication adherence reminders.
  Arms: Intervention

SUMMARY:
This study aims to conduct a 12-month randomized controlled trial to adapt the mobile app, WiseApp, and a smart pill dispenser for Spanish-speaking people living with HIV (PLWH) in the New York City (NYC) area and La Romana, Dominican Republic (DR). The study will assess the efficacy and sustainability of WiseApp as well as identify barriers with its widespread use among Spanish speakers. With disproportionately high rates of HIV in the New York City area and the Dominican Republic, this project seeks to identify distinct contextual factors related to Spanish speaking people living with HIV and increase the likelihood of engagement with technology and improvements in clinical outcomes.

DETAILED DESCRIPTION:
While efforts have been made, deficits remain in antiretroviral therapy (ART) adherence and viral suppression among PLWH. There are gaps in HIV treatment success that are particularly present in racial and ethnic minority populations, especially among Latinos in the Northeast United States (US) and the Caribbean. The progression and premature deaths among PLWH have been attributed to insufficient engagement in medical care and adherence to HIV treatments. Access and adherence to ART are important to therapeutic success and help determine long-term health outcomes in PLWH. The investigators studied racial/ethnic minorities and their providers to identify the impact a mobile app can have to improve health outcomes. The Agency for Healthcare Research and Quality (AHRQ) helped create this app and integrated it with a smart pill box (CleverCap) which allows PLWH to monitor their medication adherence. The tool, WiseApp, is a better method than other ART adherence methods because the app is linked to the smart pill box and is currently being evaluated in random-control trials (RCT) in New York City. There is also a need to develop and test self-management interventions for Spanish speaking Latino PLWH because they are the largest and fastest growing ethnic minority group in the US and are disproportionately affected by HIV. The investigators suggest the transfer of WiseApp to Latinos in the US and the DR by translating it to Spanish and making it culturally accessible. The project will use health information technology to facilitate the collection of medication adherence, quality of life, and symptom burden data.

This study aims to adapt WiseApp for Spanish speaking PLWH and conduct RCT to assess the app's efficacy and sustainability. The study will identify barriers and facilitators to the widespread use of the app and builds on the strong linkage between Columbia University and Clínica de Familia in the DR. This project is also enhanced by utilizing the strong presence of Latinos in the Washington Heights neighborhood of NYC, the disproportionately high rates of HIV in the DR, and patterns of movement of people between NYC and the DR. Additionally, the study focuses on AHRQ priority populations such as chronically ill, inner-city, low-income, and racial/ethnic minority persons.

ELIGIBILITY:
Inclusion Criteria:

* Able to speak, read, and write in Spanish;
* Aged ≥18 years;
* Willing to participate in any assigned arm of the intervention;
* Have an HIV-1 RNA level >50 copies/mL;
* Own a smartphone (DR participants who are eligible but without access to a smartphone will get one as part of the study at the time of enrollment); and
* Ability and willingness to provide informed consent for study participation and consent for access to medical records.

Exclusion Criteria:

* Reside in a nursing home, prison, and/or receiving in-patient psychiatric care at time of enrollment;
* Terminal illness with life expectancy <6 months;
* Planning to move out of the area in the next 12 months;
* A cognitive state minimum score measured by the Mini-Mental State Examination (MMSE) to ensure participants are oriented to time and place.
* Spouses/partners may not enroll in this study. The study will be limited to only 1 person from the same family/domestic household.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 248 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Change in self-reported ART adherence | Baseline, 3 month follow up, 6 month follow up, and 12 month follow up
  Self-reported ART adherence is a single-item self-report measure on a linear scale of 0-100 with zero indicating lowest adherence and 100 indicating highest adherence.

SECONDARY OUTCOMES:
Change in cluster of differentiation 4 (CD4) Count | Baseline, 3 month follow up, and 6 month follow up
  Using blood samples obtained during study visits, CD4 count will be used to assess ART adherence.
Change in Viral Load | Baseline, 3 month follow up, 6 month follow up, and 12 month follow up
  Using blood samples obtained during study visits, viral load levels will be used to assess ART adherence.
Change In Participant's Self-reported Health-related Quality of Life Score | Baseline and 12 month follow up
  Health-related quality of life will be measured with the Patient-Reported Outcomes Measurement Information System® (PROMIS)-29 measure, which measures 7 domains of health-related quality of life with 4 questions in each section pertaining to how that participant's health influences their life. In general, each question has five response options ranging in values from 1-5. To find the total raw score for this form with all the questions answered, the values from the responses of each question are summed. Raw scores are then translated into a T-score for each participant, which rescales the raw score into a standardized T-score with a mean of 50 and standard deviation (SD) of 10. Consequently, a person with a T-score of 40 would be one SD below the mean.

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Schnall, PhD, MPH, Principal Investigator — Columbia University
Locations (2):
- Columbia University Irving Medical Center, New York, New York, United States
- Clinica de Familia La Romana, La Romana, Dominican Republic, Dominican Republic

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Olaya F, Brin M, Caraballo PB, Halpern M, Jia H, Ramirez SO, Padilla JJ, Stonbraker S, Schnall R. A randomized controlled trial of the dissemination of an mHealth intervention for improving health outcomes: the WiseApp for Spanish-speakers living with HIV study protocol. BMC Public Health. 2024 Jan 17;24(1):201. doi: 10.1186/s12889-023-17538-y. PMID 38233908